CLINICAL TRIAL: NCT04128631
Title: Role of of F-18-fluoro-deoxy-glucose (FDG) PET/CT in Thyroid Cancer Patients With Negative I-131whole Body Scan and Elevated Thyroglobulin Level or Positive Anti Thyroglobulin Antibodies
Brief Title: Thyroid Cancer and (FDG)PET/CT Scan
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, RMFarghali, Principal investigator, Assiut University
Other Study IDs: FDGPET
Record Dates: First submitted 2019-09-26; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-09

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PET/CT: group of patients will do F-18FDG PET/CT scan after negative whole body scan with elevated serum thyroglobulin Antibody or Thyroglobulin levels.

SUMMARY:
Background and Rational

(Introduction)

Differentiated thyroid carcinoma (DTC) have favorable prognosis. Overall 10-year survival is 93% for papillary carcinoma, and 85% for follicular carcinoma(1). After total thyroidectomy followed by radioiodine remnant ablation, DTC patients are screened for recurrence by measuring the levels of both Tg and TgAb and I-131 whole body scan (WBS) in the follow-up (2) It is reported that elevated TgAb may indicate the recurrent and/or metastatic disease and can be used as an alternative of the tumor marker for DTC . The I-131 WBS has high specificity to detect recurrence (50 to 60% in papillary thyroid carcinoma and 64 to 67% in follicular thyroid carcinoma) (3,4). The I-131WBS showed negative finding in 10 to 15% of patients with detectable serum Tg levels(5). Two factors may account for discrepancy between serum Tg and I-131 WBS . First, the tumor size might be too small to be detected by WBS. Second, the tumor cell may lose the ability to trap radioiodine while still able to secret Tg(6,7). It becomes necessary to investigate with other modalities to identify possible residual disease to initiate the appropriate treatment. (8)

Positron emission tomography with 2-deoxy-2-[fluorine-18]fluoro- D-glucose integrated with computed tomography (18F-FDG PET/CT) has emerged as a powerful imaging tool for the detection of various cancers. (9)

The combined acquisition of PET and CT has synergistic advantages over PET or CT alone and minimizes their individual limitations. (10)

It is a valuable tool for staging and re staging of some tumors and has an important role in the detection of recurrence in asymptomatic patients with rising tumor marker levels and patients with negative or equivocal findings on conventional imaging techniques.(11)

Aim of the study

The aim of this study was to evaluate the diagnostic accuracy of (PET/CT) in patients with suspected thyroid cancer recurrence or metastasis , with differentiated thyroid cancer (DTC) patients who show elevated serum thyroglobulin (Tg) or antithyroglobulin antibody (TgAb) level with negative radioiodine whole body scan (I-WBS).

DETAILED DESCRIPTION:
Design and Methodology

Study design:-

It's a prospective study for the group of patients who will do F-18FDG PET/CT scan after negative whole body scan with elevated serum thyroglobulin Antibody or Thyroglobulin levels.

Pre-study investigations:-

* All patients at this study should have histopathological evidence of DTC
* serum TSH level
* serum TG & antiTG antibodies levels
* radioactiveiodine whole body scan (I-WBS)
* Neck ultrasound
* Blood glucose level

Radioisotopes:

Iodine-131 (I-131) is an important radioisotope of iodine as a major product of Uranium fission. It is a β-emitting radionuclide with a maximum energy of 606 keV and an average energy of 191 keV. Average range of β-particles in tissue is 0.8 mm and has a principal γ-ray of 364 keV. It has a radioactive decay half-life of about eight days. Only well-differentiated thyroid cancer cells concentrate radioiodine to a significant degree.

F-18-fluoro-2-deoxyglucose (FDG) is a positron emitting radiotracer that is transported intracellularly and phosphorylated by hexokinase to FDG-6-PO4 through the same cellular membrane transport pathways as glucose. Unlike glucose, however, FDG-6-PO4 is subsequently trapped intracellularly due to lack of further metabolism from insufficient amounts of glucose phosphatase. After intravenous administration, this substrate accumulates in tumors during the uptake phase, and whole body imaging can then be performed to identify regions of high glycolytic activity. and can be used to characterize and localize many types of tumors as well as determining stage and sites of recurrent disease.

Patient preparation

* Patients fasted for at least 6 hours before F-18FDG PET/CT imaging with the exception of water intake.
* The blood glucose level was measured before tracer injection. The blood glucose levels of all patients should be less than 150 mg/dL .
* An intravenous catheter was placed for radiopharmaceutical administration,
* After tracer injection, the patients rested on a comfortable chair during the 18F-FDG uptake period

F-18FDG PET/CT Imaging

PET/CT was initiated (45-60) min after injection of the F-18-FDG, Each patient received 400-610 MBq (11-16.5 mCi) of 18F-FDG intravenously. CT was performed before acquisition of the PET data in a single step with the patients supine. First, a scout scan was obtained to determine the axial range of the study. The scanning parameters for whole-body CT craniocaudal scanning are 130 kV, 80-120 mAs, 5-mm collimation, and a pitch of 1.6. During the scan, patients have to maintain shallow respiration.

The subsequent 3-dimensional PET data acquisition included 4-6 bed positions, (4 min per bed position) over the same axial extent. The PET acquisition included a dead time correction and online delayed coincidence subtraction to correct for random coincidences. Rescaled CT images were used to produce attenuation correction values for the PET emission reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* · This study will include thyroid cancer patients of wide age ranges, who underwent total thyroidectomy with negative radioactive iodine whole body scan (I-WBS) and elevated stimulated thyroglobulin (sTg) or thyroglobulin antibody (TgAb) levels.

  * Patients able to sleep in a fixed position for 20 minutes.

Exclusion Criteria:

Patients unable to sit calm without movement during imaging.

* Severely ill patients.
* Patients' blood glucose &GT; 11.1 mmol/L (200 mg/dL) measured by glucometer immediately prior to scan.
* Pregnancy

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include thyroid cancer patients of wide age ranges, who underwent total thyroidectomy with negative radioactive iodine whole body scan (I-WBS) and elevated stimulated thyroglobulin (sTg) or thyroglobulin antibody (TgAb) levels.
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2019-10-30 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence and metastasis | six months
  Detection of recurrence or metastasis in patient with negative radioactive iodine scan and elevated stimulated thyroglobulin (sTg) or thyroglobulin antibody (TgAb) levels.By progressively increase level of serum Thyroglobulin or thyroglobulin antibodies

SECONDARY OUTCOMES:
Improve survival rate | six months
  initiate appropriate treatment to those patients improve survival and quality of life